CLINICAL TRIAL: NCT01399151
Title: Assessment of Vitamin D Supplementation and Immune Function
Acronym: FL-82
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: WHNRC 213949-1; USDA CRIS 5306-51530-018-00D (Other Grant/Funding Number: USDA)
Record Dates: First submitted 2011-06-30; First posted 2011-07-21 (Estimated); Last update posted 2014-04-22 (Estimated); Status verified 2014-04

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D; Immune function
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Vitamin D - Treatment 1 (Experimental): 400 IU/day Vitamin D
  Interventions: Dietary Supplement: Vitamin D - Treatment 1
- Vitamin D- Treatment 2 (Experimental): 2,000 IU/day Vitamin D
  Interventions: Dietary Supplement: Vitamin D - Treatment 2
- Vitamin D- Treatment 3 (Experimental): 5,000 IU/day Vitamin D
  Interventions: Dietary Supplement: Vitamin D - Treatment 3

INTERVENTIONS:
Dietary Supplement: Vitamin D - Treatment 1 — Volunteers will take a 400 IU/day dose of Vitamin D for 12 weeks.
  Arms: Vitamin D - Treatment 1
Dietary Supplement: Vitamin D - Treatment 2 — Volunteers will take a 2,000 IU/day dose of Vitamin D for 12 weeks.
  Arms: Vitamin D- Treatment 2
Dietary Supplement: Vitamin D - Treatment 3 — Volunteers will take a 5,000 IU/day dose of Vitamin D for 12 weeks.
  Arms: Vitamin D- Treatment 3

SUMMARY:
Hypothesis:

Volunteers with vitamin D insufficiency (serum 25(OH)D 25-50 nmol/L) given intermediate or high dose vitamin D supplements (2,000 or 5,000 IU per day) will have increased production of anti-bacterial peptides and interleukin-1, decreased production of other pro-inflammatory cytokines, increased production of regulatory cytokines and an enhanced T- and B-cell response to a tetanus vaccine compared to vitamin D insufficient subjects given low dose vitamin D supplements (400 IU per day).

DETAILED DESCRIPTION:
Specific Aim 1:

Determine if high dose vitamin D supplements decrease the production of proinflammatory and increase the production of regulatory cytokines and chemokines by innate immune cells stimulated ex vivo.

Specific Aim 2:

Determine if high dose vitamin D supplements decrease serum markers of inflammation and increase serum and cellular levels of defensive molecules (e.g., cathelicidin).

Specific Aim 3:

Determine if high dose vitamin D supplements decrease blood levels of proinflammatory T-helper type 1 (Th1) and Th17 cells and increase levels of anti-inflammatory T-regulatory (Treg) and Th2 cells.

Specific Aim 4:

Determine if high dose vitamin D supplements increase antigen specific T cell and B cell responses after tetanus vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-49 (men) and 20-45 (women)
* BMI 18.5-30
* Serum 25OH Vitamin D 25-50 nmol/L

Exclusion Criteria:

* Pregnant or nursing women
* Daily smoker
* Anemia (Hgb<12 mg/dL for women and <13 mg/dL for men) determined at initial visit
* Any report or diagnosis of disease or chronic condition that may affect vitamin D absorption such as cystic fibrosis, celiac disease, surgical removal of part of the stomach or intestines, and some forms of liver disease
* Diagnosis of hyper parathyroidism and chronic granulomatous disease, which increases risk of hypercalcemia.
* Planned to travel to a location at which either altitude or latitude would result in significant vitamin D synthesis during the study period.
* Not previously vaccinated with TT, or vaccinated within five years
* Use of steroids or antibiotics within the past 4 weeks
* Current use of nutritional supplements that may alter immune function such as omega 3 fatty acid supplements
* Current use of anti-inflammatory or anti-convulsion medications
* Self reported history of significant adverse response to previous vaccinations

Ages: 20 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2011-01; Primary Completion 2013-12 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change in Cathelicidin levels in granulocytes | 0, 8, and 12 weeks
Change in cytokine levels from stimulated Periferal Blood Mononuclear Cells | 0, 8 and 12 weeks
Change in serum cytokines and acute phase proteins | 0, 8 and 12 weeks
Change in markers of response to tetanus vaccination | 0, 8, 9, 10 and 12 weeks
  Markers of response to tetanus vaccine include tetanus-specific proliferation and production of cytokines by CD4 T-helper cells.
Change in serum 25OH Vitamin D | 0, 4, 8, and 12 weeks
Change in urinary calcium-to-creatinine ratio | 0, 2, 4, 6, 8 and 10 weeks

SECONDARY OUTCOMES:
Change in level of 5-lipoxygenase protein in granulocytes | 0, 8 and 12 weeks
Change in production of leukotrienes in granulocytes | 0, 8, and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Charles Stephensen, PhD, Principal Investigator — WHNRC, ARS, University of California Davis
Locations (1):
- Western Human Nutrition Center, University of California Davis, Davis, California, United States

REFERENCES:
- See also: USDA Western Human Nutrition Research Center — http://www.ars.usda.gov/Main/docs.htm?docid=11240